CLINICAL TRIAL: NCT05451563
Title: Double-S: a Wearable Device for Erectile Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael Eisenberg, Michael Eisenberg M.D., Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 65457
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Double-S arm (Experimental): Participants will be asked to use the wearable penile device during intercourse.
  Interventions: Device: Double-S

INTERVENTIONS:
Device: Double-S — Wearable device for intercourse

SUMMARY:
The purpose of this study is to use a minimally invasive erectile device for patients suffering from erectile dysfunction.

DETAILED DESCRIPTION:
The purpose of the study is to use a minimally invasive erectile device support to provide to patients suffering from erectile dysfunction the possibility to achieve satisfactory penetrating intercourse.

The goal of this is to help men who have issues with erectile function (e.g.after radical prostatectomy for prostate cancer, vascular or metabolic erectile dysfunction non-responsive to phosphodiesterase-5 inhibitor medications, etc.) to have medication-free mechanical support for their penis in order to obtain sexual penetration satisfactorily.

ELIGIBILITY:
Inclusion Criteria:

* males >18 years old suffering from any cause moderate to severe erectile dysfunction (e.g. ED after radical prostatectomy and/or radiation therapy for prostate cancer and or other pelvic malignancies affecting the sexual potency; emotional and psychological ED; organic vascular and/or metabolic ED etc.)
* having a female partner willing to participate in the study

Exclusion Criteria:

* not willing to attempt sexual vaginal intercourse with their partner
* inability to wear/operate the external penile device for any reason

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in modified International Index of Erectile Dysfunction score | baseline and up to 1 month post-baseline
  score 0 to 30 with higher score meaning better erectile function

CONTACTS AND LOCATIONS:
Overall Officials: Michael Eisenberg, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Healthcare, Stanford Hospital, Stanford, California, United States